CLINICAL TRIAL: NCT04946955
Title: Intervention Research for Suicide Prevention Among Adolescents and Young Adults in the General Population Using E-health Tools and a Promotion System Involving the Civilian Population
Brief Title: Adaptation of a French E-health Tool for Suicide Prevention in Young Populations
Acronym: E-psYouth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180676
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-06

CONDITIONS: Suicide; Depression; Psychological Distress; Anxiety Disorders
Keywords: Primary care; Prevention; Suicide; Mental health; Young adults; Adolescents
MeSH Terms: conditions — Suicide; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Within the framework of the project, the beneficiary public is the population of young adults and adolescents between 11 and 25 years old likely to connect to a mobile application and an associated website dedicated to the prevention of psychological suffering and suicide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application and website with promotion (Experimental): Development of an application and a website to de-stigmatise mental health and support the user in seeking help
  Interventions: Other: Application and website with or without promotion
- Application and website without promotion (Other)
  Interventions: Other: Application and website with or without promotion

INTERVENTIONS:
Other: Application and website with or without promotion — Development of an application and a website to de-stigmatise mental health and support the user in seeking help

SUMMARY:
"France's suicide rate is among the highest in Europe, with the young among the more at risk. Several European projects have demonstrated the effectiveness of using e-tools in suicide prevention particularly for hard-to-reach populations.

Lessons from StopBlues, an e-health tool (application/website) for suicide prevention in the general population developed in 2018 which was promoted by municipalities and general practitioners, show the necessity to adapt its content for young people.

The objective is to develop an e-health tool for suicide prevention targeting adolescents and young adults with psychological pain by adapting StopBlues and its promotional plan.

The detailed content of the e-health tool and its promotional plan will be determined via a literature review followed by individual and group interviews with experts and youth, with StopBlues as a starting part.

This adaptation of StopBlues will allow to reach a larger audience by offering a more suitable solution for this vulnerable population. A web-portal will serve as an entry point for both StopBlues and the new e-tool where users will be redirected to one of the tools/modules according to their profile and respective needs. "

DETAILED DESCRIPTION:
"Context: France's suicide rate is among the highest in Europe, with the young among the more at risk. Several European projects have demonstrated the effectiveness of using e-tools in suicide prevention particularly for hard-to-reach populations.

Lessons from StopBlues, an e-health tool (application/website) for suicide prevention in the general population developed in 2018 which was promoted by municipalities and general practitioners, show the necessity to adapt its content for young people.

Research objectives:

Phase I: Development of the e-health tool The objective of this part is to set up a consultation to co-construct, on the one hand, an e-mental health tool including a smartphone application and its website with and for young people adapted to their age group and, on the other hand, the promotionnal plan.

Methodology: The detailed content of the e-health tool and the promotional tools will be determinated with a literature review and consultations of youth and experts. Then, the investigators will rely on different networks to invite young people to an online consultation according to their age group to participate from the start to this intervention. Several means will be mobilised to involve them. the investigators will discuss with them: their feelings about the existing StopBlues adult tool (www.stopblues.fr), their perception of the specific topics that need to be addressed regarding the causes of psychological suffering, the possible solutions, the identification of speakers who act out situations that young people can identify with, their opinion on the graphic charter and design, and finally the means of dissemination that we could use to promote this tool.

The investigators will use the data saturation method to stop recruiting. The data collection necessary for the co-construction will be realised on digital platforms through surveys including questionnaires with either open questions or multiple-choice questions. The data will then be analysed using qualitative and quantitative methods.

The investigators will also use the digital platforms mobilised for this consultation to present the results and validate with participating youth the final version of the content, structure and ergonomics of the tool to be developed.

Expected results: This consultation will allow the project team to co-construct with young people an e-health intervention involving a mobile application, a website and their promotion.

The investigators also expect it to provide more precise information on:

* youth feelings about the adult version of the tool (StopBlues): its content, its ergonomics and the means of communication used (videos of professionals and testimonies);
* youth perception of the specific topics that need to be addressed regarding the causes of psychological suffering and possible solutions;
* youth opinions concerning the graphic charter, the name and logo of the tool; - and identification of some witnesses or witnesses' relatives to interview.

Phase II: Implementation of the intervention

The main objective is to assess the effectiveness in reducing suicidal acts of a suicide prevention program for young adults in the general population, combining an e-health tool and its promotion by local authorities. The secondary objectives are to assess the effect of the programme on youth in terms of :

* efficiency of the programme and its total and sectoral budgetary impact.
* quality of life
* mental health status (anxiety and depressive symptoms, addictions, eating disorders, suicide risk)
* use of formal and informal help
* depression detected by a relative
* user satisfaction
* effectiveness of the promotion on the intensity of use of the e-health tool
* completion of the safety plan
* school or employment integration
* effectiveness of the tool according to the social status of users
* spillover effect of the programme on the youth suicide prevention policy: measures put in place secondarily by the communities involved
* the process of implementation of the promotion by the communities
* barriers and levers for studying transferability. Methodology: The trial will last 18 months from the moment the e-tool will be online. Data will be collected both from health data bases and at the individual user level.

Expected results: The intervention, which includes the development of an e-health tool for young people and its implementation with a promotion, will make it possible to confirm the applicability of the intervention model used for adults for suicide prevention in the general population (StopBlues), on a more restricted population (the E-psyjeunes tool), that of 11-25 year olds. This project will make it possible to address the question, mentioned many times when StopBlues was set up, of psychological suffering of young people. The malaise of adolescents and young adults is unique and requires specific development. Through this project, a response can be provided to the many actors (young people, associations, health professionals, local authorities, etc.) looking for help and solutions.

The investigators believe that this intervention will lead to a reduction in suicidal acts (suicides and attempted suicides) of young people. With the use of these tool, users should develop a better knowledge of mental health and suicide in general, but also of their own mental health status. They should also become more aware of the formal and informal ways of seeking help and their use of help should increase, as well as their actions increasing well-being/coping strategies implementation. A decrease in the stigma of mental disorders is also expected among young people."

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for users in the study were adolescents and young adults:

* between 11 and 25 years old
* living in France
* with a valid email account and internet access
* volunteers
* no objection from the legal representative for minors.

The criterion for non-inclusion will be the refusal of the users and/or the legal representative for minors to participate."

Exclusion Criteria:

-

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12000000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
number of suicidal acts (completed suicide and suicide attempts) | 12 month
  The number of completed suicides will be extracted from the database of the Epidemiology center on medical causes of deaths (CépiDc) for each local authority participating. The number of attempted suicides will be extracted from the national database of public and private hospital admissions (PMSI-MCO) and the national emergency database (Oscour).

CONTACTS AND LOCATIONS:
Overall Officials: Karine Chevreul, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- ASSISTANCE PUBLIQUE HOPITAUX DE PARIS (URC Eco, Hôpital Hôtel-Dieu), Paris, France

IPD SHARING:
Plan to Share IPD: No